CLINICAL TRIAL: NCT02321878
Title: Post-marketing Surveillance (Special Use-results Surveillance) on Use With Liraglutide (Victoza®)
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN2211-4175; U1111-1157-6701 (Other: WHO)
Record Dates: First submitted 2014-12-17; First posted 2014-12-22 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Liraglutide
  Interventions: Drug: liraglutide

INTERVENTIONS:
Drug: liraglutide — Liraglutide (Victoza®) will be prescribed by the physician under normal clinical practice conditions.
  No treatment given.

SUMMARY:
This trial is conducted in Asia. The aim of this trial is to evaluate safety and effectiveness of Victoza® in patients with type 2 diabetes mellitus (T2DM) in combination with antidiabetes agents other than sulfonylurea under post-marketing normal clinical practice conditions.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any study-related activities (Study-related activities are any procedure related to recording of data according to the protocol)
* Patients with T2DM (type 2 diabetes mellitus) who the physician has decided to start treatment with Victoza® in combination with insulin or OAD (oral anti-diabetes drug) other than SU (sulfonylurea)
* Male or female, no age limitation

Exclusion Criteria:

* Previous participation in this study or NN2211-3772 Participation is defined as informed consent obtained for this study or enrolment for NN2211-3772
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation
* Patients who are on Victoza® or have previously been on Victoza® within 3 month before the enrolment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male or female patients with T2DM who the physician has decided to start on treatment with Victoza® in combination with insulin or oral anti-diabetes drug (OAD) other than SU (Sulfonylurea) will be eligible for this study.
Sampling Method: Non-Probability Sample
Enrollment: 1092 (Actual)
Dates: Start 2014-12-15 (Actual); Primary Completion 2017-06-16 (Actual); Study Completion 2017-06-16 (Actual)

PRIMARY OUTCOMES:
Number of AEs (adverse events) | Week 0-52

SECONDARY OUTCOMES:
Number of adverse reactions (ARs) | Week 0-52
Change in HbA1c (glycosylated haemoglobin) | Week 0, week 52

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (5):
- Japan (5):
  - Novo Nordisk Investigational Site, Chichibu
  - Novo Nordisk Investigational Site, Koriyama-shi, Fukushima
  - Novo Nordisk Investigational Site, Oyama-shi, Tochigi
  - Novo Nordisk Investigational Site, Tagajō-shi
  - Novo Nordisk Investigational Site, Tokyo

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com